CLINICAL TRIAL: NCT01973400
Title: A Clinical Study on the Neuroprotection by Tocotrienols in Type 1 and Type 2 Diabetes Mellitus
Brief Title: Neuroprotection by Tocotrienols in Type 1 and Type 2 Diabetes Mellitus
Acronym: VENUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Clinical Research Centre, Malaysia (Other); Malaysia Palm Oil Board (Other Government)
Responsible Party: Principal Investigator, Yuen Kah Hay, Professor Dr., Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: VENUS-7327; NMRR-10-948-7327 (Registry Identifier: National Medical Research Register (Malaysia))
Record Dates: First submitted 2013-10-24; First posted 2013-10-31 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Diabetic Neuropathy; Cognitive Impairment
MeSH Terms: conditions — Diabetic Neuropathies; Cognitive Dysfunction | interventions — Tocotrienols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tocotrienol (Experimental): 200 mg, twice a day, 12 months
  Interventions: Dietary Supplement: Tocotrienol
- Placebo (Placebo Comparator): 200 mg, twice a day, 12 months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Tocotrienol — Palm-Oil derived Vitamin E, tocotrienol
  Arms: Tocotrienol
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Given that the tocotrienols have been shown to possess neuroprotective effects and that both type 1 and type 2 diabetes can lead to peripheral neuropathy and cognitive impairment, the present study aims to determine the beneficial effects of tocotrienols in ameliorating such neurological related events in both type 1 and type 2 diabetic patients.

DETAILED DESCRIPTION:
Neuropathy affects approximately 30-50% of all diabetic patients and is the commonest form of neuropathy in the developed world. Pain is the most distressing symptom of neuropathy and the main factor that prompts the patient to seek medical advice. About 16-26% of diabetes patients experience chronic neuropathic pain. An animal study revealed that treating rats with α-tocopherol and tocotrienol for 10 weeks significantly improved all the biochemical and behavioral outcomes of alcohol-induced neuropathy in a dose-dependent manner with more potent effects observed with tocotrienols. The study demonstrates the effectiveness of tocotrienols in attenuation of alcoholic neuropathy.

Cognitive dysfunction is a less addressed and not as well recognized complication of diabetes. Patients with type 1 and type 2 diabetes mellitus have been found to have cognitive deficits that can be attributed to their disease. Both old age and diabetes are independently associated with an increased risk of cognitive dysfunction; the risk is even greater for older adults with diabetes. Cognitive Function is the term used to describe a person's state of consciousness (alertness and orientation), memory, and attention span. It has been suggested that Vitamin E, including tocopherols and tocotrienols, can help to improve cognitive function and stall cognitive decline through its antioxidant effects. A reason for this nutrient's success at preventing oxidative damage in brain cells is its fat-soluble criteria. During the World Alzheimer's Congress held in July 2001, it was reported that high intakes of vitamin E effectively lessened memory loss and cognitive dysfunction among more than 6,000 elderly subjects who were generally taking Vitamin E between 200 to 400 IU per day.

Tocotrienols, in particular α-tocotrienol have been shown to possess neuroprotective effect independent of anti-oxidant activity. Using cell-based studies, α-tocotrienol but not α-tocopherol was shown to prevent glutamate-induced neuronal cell death at nanomolar concentrations. Later studies showed that α-tocotrienol conferred protection against glutamate and stroke-induced neurodegeneration in rats.

In view of the above neuroprotective property of tocotrienols, researchers have proceeded to demonstrate that tocotrienols supplementation helped to reverse neuropathic pain in diabetic rats. It has been postulated the beneficial properties of tocotrienols are due to their suppressive effects on the oxidative-nitrosative stress, inflammatory cytokine release and caspase-3 which are implicated in the pathogenesis of diabetic neuropathy.

In the same year, tocotrienols were shown to prevent cognitive deficits and attenuate alcoholic peripheral neuropathy associated with selective neuronal damage due to chronic alcohol consumption. Moreover, the beneficial effects were found to be more pronounced with tocotrienols compared to tocopherols. It has been postulated that the anti-oxidants property of tocotrienols, the suppression of nitrosative stress and elevated cytokines levels together with acetylcholinesterase activity in the brain regions contributes significantly in preventing the chronic alcohol-induced cognitive deficits in rats.

Yuen and his group are currently conducting a clinical study in human subjects on neuroprotective effects of tocotrienols (NCT00753532). In the study, subjects were followed up for 2 years to determine the volume of white matter lesions on repeated MRI after treatment with tocotrienol as compared to placebo. White matter lesions are related to vascular events in the brain and represent subclinical infarcts, resulting in death/ degeneration of neurons and are positively correlated to cognitive impairment. Preliminary results from an interim analysis are encouraging; patients on tocotrienols shown significant reduction in volume of white matter lesion (confidential communication).

ELIGIBILITY:
Inclusion Criteria:

* Diabetic adults ( both type 1 or 2) ≥20 years old with diabetic peripheral neuropathy with Total Symptom Score(TSS) ≥ 3 points.
* Patients with type 1 diabetes (duration of ≥5 years).
* Patients with type 2 diabetes (at diagnosis).
* Patients with Neuropathy Impairment Score(NIS) > 2

Exclusion Criteria:

* Patients HbA1c >12%.
* Patients with hypoglycemia or conscious impairment at the time of test conduction.
* Patients exhibiting symptoms of peripheral vascular disease with absence of 2 foot pulses on the same foot (Posterior tibialis, Dorsalis pedis)
* Immuno-compromised patients.
* Patients with severe visual impairment, history of psychosis; schizophrenia; bipolar disorder; current depression or brain trauma and patients with alcohol dependence or drug abuse such as cocaine, heroin, etc.
* Those having lesions with a propensity to bleed (e.g., bleeding peptic ulcers), those having a history of hemorrhagic stroke and those with inherited bleeding disorders (e.g., hemophilia) or patients on warfarin.
* Pregnancy and lactation.
* Patients with renal function test of more than 150 umol/L (serum creatinine).
* Patients with liver function test of more than 5 times of the upper normal range
* Active infection or infectious diseases.
* Other significant uncontrolled medical illnesses that may interfere with drug administration or interpretation of results.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-06; Primary Completion 2015-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Total Symptoms Score (TSS) (pain, paresthesia, burning, and numbness)of patients with diabetes type 1 and 2 neuropathy. | 1 year

SECONDARY OUTCOMES:
Neuropathy Impairment Score (NIS) of patients with diabetes type 1 and 2 neuropathy | 1 year

OTHER OUTCOMES:
Mini Mental State Examination (MMSE) score, Montreal Cognitive Assessment (MoCA) test. | 1 year
  Measures the effects of tocotrienols on cognitive impairment in type 1 and type 2 diabetes mellitus

CONTACTS AND LOCATIONS:
Overall Officials: Kah Hay Yuen, PhD, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Seberang Jaya Hospital, Seberang Jaya, Pulau Pinang, Malaysia

REFERENCES:
- [Derived] Vitamin E in Neuroprotection Study (VENUS) Investigators; Hor CP, Fung WY, Ang HA, Lim SC, Kam LY, Sim SW, Lim LH, Choon WY, Wong JW, Ch'ng ASH, Beh KKM, Wee HC, Ong LM, Khan NAK, Sulaiman SAS, Shuaib IL, Bakar A, Yusof Y, Yusof YM, Abu Bakar F, Tang WS, Teh HL, Wahid NA, Saaidin S, Idris N, Yoon CK, Ong HN, Ganapathy JT, Loo CE, Samy MM, Zainal H, Dharan SCS, Ooi BY, Teoh PY, Tye YL, Yeoh CA, Low DW, Looi I, Yuen KH. Efficacy of Oral Mixed Tocotrienols in Diabetic Peripheral Neuropathy: A Randomized Clinical Trial. JAMA Neurol. 2018 Apr 1;75(4):444-452. doi: 10.1001/jamaneurol.2017.4609. PMID 29379943